CLINICAL TRIAL: NCT02499731
Title: Strong Hearts, Healthy Communities: A Rural Community CVD Prevention Program
Brief Title: Strong Hearts: Rural CVD Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Montana State University (Other); Tufts University (Other); Bassett Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB #: 1402004505
Record Dates: First submitted 2015-07-01; First posted 2015-07-16 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Heart Disease; Cardiovascular Disease; Sedentary Lifestyle; Overweight; Obesity
Keywords: physical activity; nutrition; social network
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Sedentary Behavior; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strong Hearts, Healthy Communities (Experimental): Full Intervention participants will meet twice per week for one hour each time, for approximately 6 months plus monthly community meetings and events. Participants will learn and practice good nutrition and physical activity for improved individual, family and community health.
  Interventions: Behavioral: Strong Hearts, Healthy Communities
- Strong Hearts, Healthy Women (Experimental): Strong Hearts, Healthy Women minimum intervention participants meet once per month for an hour each time for 6 months. Participants will learn and discuss techniques and strategies to improve personal health.
  Interventions: Behavioral: Strong Hearts, Healthy Women

INTERVENTIONS:
Behavioral: Strong Hearts, Healthy Communities — We will evaluate the efficacy of the SHHC curriculum in a 24-week community-based randomized controlled intervention trial. We will compare changes in CVD-related anthropometric, physiologic, behavioral, and psychosocial parameters between subjects in 8 intervention and 8 control communities. In addition, we will evaluate changes in behavior, attitudes, and knowledge among SHHC intervention subjects' "social network".
  Other Names: Strong Hearts for Montana; Full intervention
  Arms: Strong Hearts, Healthy Communities
Behavioral: Strong Hearts, Healthy Women — The Strong Hearts, Healthy Women (minimal intervention) will meet once per month for an hour each time for 6 months.
  Participants will learn and discuss techniques and strategies to improve personal health.
  Other Names: Strong Hearts for Montana; Minimal intervention
  Arms: Strong Hearts, Healthy Women

SUMMARY:
Strong Hearts, Healthy Communities is a research study which aims to reduce cardiovascular disease (CVD), improve quality of life, and reduce CVD related health care costs in rural communities.

The investigators' aim is to better understand how changes in lifestyle can affect the health of rural women and others in their communities.

DETAILED DESCRIPTION:
There are notable cardiovascular disease (CVD) disparities among people living in rural settings, particularly medically underserved rural areas. Complex factors such as socioeconomic disadvantage, social and cultural dynamics, geographic distances/barriers, and limited access to healthcare, healthy foods, and/or physical activity opportunities contribute to the issue. The objective of Strong Hearts, Healthy Communities (SHHC) is to reduce rural CVD disparities through civic engagement and implementation of a community-based intervention in 16 underserved rural towns. In Montana, SHHC builds upon a long-standing collaboration with National Institute of Food and Agriculture cooperative extension educators, who will implement the project. SHHC in New York will work with a health care system to implement the project. There is limited knowledge about how programs and services can move beyond commonly used individual-level approaches-which have limitations in terms of cost, impact, reach, and sustainability-to effectively reduce rural CVD health disparities using an integrated, multi-level, community-engaged approach. The objective of Strong Hearts, Healthy Communities (SHHC) is to address this gap in knowledge and practice by working with residents, practitioners, health educators, local leadership, and other stakeholders in 16 medically underserved rural towns to develop and test a comprehensive program designed to: a) improve diet and physical activity behaviors, b) promote local built environment resources, and c) shift social norms about active living and healthy eating through civic engagement, capacity building, and community-based programming.

FORMATIVE RESEARCH (STAGE1: Completed) The investigators conducted community audits, focus groups, and key informant interviews with members of the above key groups to gather in-depth data about a number of topics related to CVD awareness and risk factors. These topics included: economic, healthcare, and social/cultural factors, as well as, barriers and facilitators to healthy eating and active living. The community audit and qualitative data gathered during the formative research, as well as, feedback from extension educators and the National Advisory Board has informed and been incorporated in the development and refinement of the SHHC curriculum.

RANDOMIZED CONTROLLED INTERVENTION (STAGE 2) In the second phase of the project, the investigators will evaluate the efficacy of the SHHC curriculum in a 24-week community based randomized controlled intervention trial. The investigators will compare changes in CVD-related anthropometric, physiologic, behavioral, and psychosocial parameters between subjects in 8 intervention and 8 control communities. In addition, the investigators will evaluate changes in behavior, attitudes, and knowledge among SHHC intervention subjects' "social network".

ELIGIBILITY:
Inclusion Criteria:

* Not currently physically active
* BMI greater than or equal to 25
* Blood pressure is less than 160/100 mm Hg
* Heart rate is between 60-100 bpm
* English-speaking
* Able and willing to obtain physician's approval to participate in either intervention
* Willing to participate in assessment activities
* Willing to make a firm commitment to participate in either intervention

Exclusion Criteria:

* Currently physically active
* Body Mass Index less than 25
* Untreated hypertension
* Heart rate lower than 60 or higher than 100 bpm
* Non-English speaking
* Not able or willing to obtain physician's approval to participate
* Not interested or willing to participate in assessment activities
* Not able or willing to make a firm commitment to participate in either intervention

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline to 6 months, 6-month follow-up, and 18-month follow-up

SECONDARY OUTCOMES:
Changes in blood pressure | Baseline to 6 months, 6-month follow-up, and 18-month follow-up
Changes in lipids | Baseline to 6 months, 6-month follow-up, and 18-month follow-up
Changes in c-reactive protein | Baseline to 6 months, 6-month follow-up, and 18-month follow-up
Changes in hemoglobin A1C | Baseline to 6 months, 6-month follow-up, and 18-month follow-up
Changes in waist circumference | Baseline to 3 months, 6 months, 6-month follow-up, and 18-month follow-up
Changes in 7-day accelerometry | Baseline to 6 months, 6-month follow-up, and 18-month follow-up
Changes in 7-day dietary recall | Baseline to 6 months, 6-month follow-up, and 18-month follow-up
Changes in healthy eating self-efficacy assessed by questionnaire | Baseline to 3 months, 6 months, 6-month follow-up, one-year follow-up, and 18-month follow-up
Changes in exercise self-efficacy assessed by questionnaire | Baseline to 3 months, 6 months, 6-month follow-up, one-year follow-up, and 18-month follow-up
Changes in healthy eating attitudes of social network of participants assessed by questionnaire | Baseline to 6 months and 6-month follow-up
Changes in exercise attitudes of social network of participants assessed by questionnaire | Baseline to 6 months and 6-month follow-up
Changes in healthy eating self-efficacy of social network of participants assessed by questionnaire | Baseline to 6 months and 6-month follow-up
Changes in exercise self-efficacy of social network of participants assessed by questionnaire | Baseline to 6 months and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Seguin, PhD, Principal Investigator — Cornell University
Locations (16):
- United States (16):
  - Broadus, Broadus, Montana
  - Chinook, Chinook, Montana
  - Choteau, Choteau, Montana
  - Columbus, Columbus, Montana
  - Forsyth, Forsyth, Montana
  - Glasgow, Glasgow, Montana
  - Harlowton, Harlowton, Montana
  - Hinsdale, Hinsdale, Montana
  - Lewistown, Lewistown, Montana
  - Plentywood, Plentywood, Montana
  - Shelby, Shelby, Montana
  - Thompson Falls, Thompson Falls, Montana
  - Cherry Valley, Cherry Valley, New York
  - Little Falls, Little Falls, New York
  - St. Johnsville, Saint Johnsville, New York
  - Sidney, Sidney, New York

REFERENCES:
- [Derived] Morgan EH, Graham ML, Marshall GA, Hanson KL, Seguin-Fowler RA. Serum carotenoids are strongly associated with dermal carotenoids but not self-reported fruit and vegetable intake among overweight and obese women. Int J Behav Nutr Phys Act. 2019 Nov 12;16(1):104. doi: 10.1186/s12966-019-0869-3. PMID 31718657
- [Derived] Folta SC, Paul L, Nelson ME, Strogatz D, Graham M, Eldridge GD, Higgins M, Wing D, Seguin-Fowler RA. Changes in diet and physical activity resulting from the Strong Hearts, Healthy Communities randomized cardiovascular disease risk reduction multilevel intervention trial. Int J Behav Nutr Phys Act. 2019 Oct 25;16(1):91. doi: 10.1186/s12966-019-0852-z. PMID 31653260
- [Derived] Wang H, Kenkel D, Graham ML, Paul LC, Folta SC, Nelson ME, Strogatz D, Seguin RA. Cost-effectiveness of a community-based cardiovascular disease prevention intervention in medically underserved rural areas. BMC Health Serv Res. 2019 May 16;19(1):315. doi: 10.1186/s12913-019-4117-y. PMID 31096977
- [Derived] Seguin RA, Paul L, Folta SC, Nelson ME, Strogatz D, Graham ML, Diffenderfer A, Eldridge G, Parry SA. Strong Hearts, Healthy Communities: A Community-Based Randomized Trial for Rural Women. Obesity (Silver Spring). 2018 May;26(5):845-853. doi: 10.1002/oby.22158. Epub 2018 Apr 10. PMID 29634086
- [Derived] Morgan EH, Graham ML, Folta SC, Seguin RA. A qualitative study of factors related to cardiometabolic risk in rural men. BMC Public Health. 2016 Apr 11;16:305. doi: 10.1186/s12889-016-2977-1. PMID 27066824
- [Derived] Seguin RA, Eldridge G, Graham ML, Folta SC, Nelson ME, Strogatz D. Strong Hearts, healthy communities: a rural community-based cardiovascular disease prevention program. BMC Public Health. 2016 Jan 28;16:86. doi: 10.1186/s12889-016-2751-4. PMID 26822982